CLINICAL TRIAL: NCT06879977
Title: Body Awareness in People With Depressive Disorder
Acronym: ABC-D
Status: Recruiting | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Christian Mittermaier, Head of Department, M.D., Johannes Kepler University of Linz
Other Study IDs: ABC-D_1
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder
Keywords: Depression; Body awareness
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with depressive disorders: Patients with depressive disorders at the beginning and end of an inpatient stay

SUMMARY:
Body awareness plays a crucial role in health and well-being. However, too little research has been carried out on how it manifests in individuals with depressive disorders. The Awareness Body Chart (ABC), a tool developed in recent years to assess body awareness, may provide new insights into the physical experience of people with depression and may lead the way in the application of body-oriented therapies in this cohort. Information about the distribution properties of the Awareness Body Chart in people with depressive disorder will be collected and analysed in this observational study.

DETAILED DESCRIPTION:
Research Questions:

* Primary Research Question What are the distribution properties of the body awareness assessed by the ABC?
* Secondary Research Questions (exploratory)

  1. Which factors (demographic, physical, psychological) correlate with body awareness?
  2. Does body awareness and mood change during an inpatient stay? Method: Observational Study Participants: 125 patients with depressive disorders at the beginning and end of an inpatient stay.

Assessments via Questionnaires:

Completion of questionnaires (partially with assistance) within the first 7 days after admission:

* Demographic data and questions about health/relevant pre-existing conditions, including body weight and height, i.e. Body Mass Index
* Awareness Body Chart (ABC)
* Like/Dislike Body Chart (L/D-BC)
* Self-Rating Mood Scale-Revised (Bf-SR)
* Simple Physical Activity Questionnaire (SIMPAQ)
* Short Form Health Survey (SF-12)
* Brief Symptom Inventory (BSI)
* Beck Depression Inventory II (BDI-II)
* Insomnia Severity Index (ISI)

Pre-Discharge Questionnaire Completion:

* ABC
* L/D-BC
* Bf-SR
* BDI-II
* ISI

Statistical Analysis:

For the analysis of the primary outcome, the ABC score for the entire sample will be presented using the mean and standard deviation or median and interquartile range, depending on the distribution properties of the ABC score. For the analysis of secondary questions, the total scores of the ABC and factor scores will be compared between men and women, between patients with and without pain, using t-tests or Mann-Whitney U-tests, and between individuals with different categories of depressive disorders or varying severities of depression using ANOVA or Kruskal-Wallis tests.

Furthermore, the correlation of body awareness with demographic data, body mass index, diagnosis group, disease duration, test results from SIMPAQ, SF-12, BSI, Bf-SR, and ISI will be investigated using correlation analyses, where the correlation coefficient will be calculated either using Pearson or Spearman, depending on the distribution of the data. Changes in body awareness and well-being during an inpatient stay will be analyzed using paired t-tests or Wilcoxon signed-rank tests.

Outlook:

The study serves as a basis for further research on body awareness in individuals with depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 69 years
* Medical diagnosis of a depressive disorder, including depressive adjustment disorder and depressive episodes in the context of bipolar disorder, i.e. one of the following ICD-10 codes:
* F32 Depressive Episode
* F33 Recurrent Depressive Disorder
* F31.3 Bipolar Affective Disorder, current mild or moderate depressive episode
* F31.4 Bipolar Affective Disorder, current severe depressive episode without psychotic symptoms
* F43.20 Adjustment Disorder with Brief Depressive Reaction
* F43.21 Adjustment Disorder with Prolonged Depressive Reaction
* Inpatient admission
* Written informed consent

Exclusion Criteria:

* Inability to fill out questionnaires with or without assistance due to language, physical, or cognitive limitations
* Acute psychotic state
* Known body schema disorders, e.g. due to significant neurological or malignant diseases, eating disorders, congenital or acquired physical limitations such as the absence of a body part
* Deafness, blindness

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with depressive disorders at the beginning and end of an inpatient stay.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Awareness Body Chart Questionnaire (ABC) | Within the first 7 days after admission
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness. In the case of pain, the pain location can also be marked on the body chart with a red pen and recorded on a 100 mm Visual Analogue Scale from 0 (no pain) to 100 (unbearable pain).

SECONDARY OUTCOMES:
Awareness Body Chart Questionnaire (ABC) | Before discharge
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness. In the case of pain, the pain location can also be marked on the body chart with a red pen and recorded on a 100 mm Visual Analogue Scale from 0 (no pain) to 100 (unbearable pain).
Like/Dislike Body Chart | Within the first 7 days after admission and before discharge
  As an extension to the ABC, this questionnaire is intended to answer the question of whether there are areas of the body that one particularly likes about oneself or that one dislikes about oneself. If yes, one can draw these with a purple color pencil ("particularly like") and/or with a gray color pencil ("do not like") in an extra Body Chart.
Self-rating mood scale - revised | Within the first 7 days after admission and before discharge
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.
Beck Depression Inventory II (BDI-II) | Within the first 7 days after admission and before discharge
  The BDI-II represents a self-rating instrument to assess the severity of depression. Four statements are given for each of 21 questions, from which the one that best describes how the person has felt in the past week is to be selected. In scoring, each item is given a score of 0 to 3, depending on the choice (higher number means higher depression scores), and after directly adding the scores of the individual items, a total score of 0 to 63 is obtained. A score of 9-13 is considered minimal depression, 14-19 is mild depression, 20-28 is moderate depression, and scores above 29 indicate severe depression.
Insomnia Severity Index (ISI) | Within the first 7 days after admission and before discharge
  The ISI is a self-assessment questionnaire used to evaluate the nature, severity, and impact of insomnia over the past two weeks. The ISI contains seven items rated with a five-point Likert scale (0 = not at all, 4 = very severe problem), with the total score ranging from 0 to 28. Higher scores indicate greater severity of insomnia. Scores from 0-7 are considered no insomnia, 8-14 is subthreshold insomnia, 15-21 is moderate insomnia, and 22-28 is severe insomnia.
Simple Physical Activity Questionnaire (SIMPAQ) | Within the first 7 days after admission
  Questionnaire to survey physical activity: It should show a snapshot of hours per day of an average day in the past week. The time in bed, the time while doing sedentary work (including dozing), while walking, while exercising and during other physical activities (such as household chores) is interrogated. The test does not measure the intensity of physical activity, but rather sorts it into the groups walking, sport and other categories.
Short Form 12 Health Survey (SF-12) | Within the first 7 days after admission
  Questionnaire on health-related quality of life. It consists of twelve questions relating to the last four weeks and yields statements about eight different dimensions of subjective health: general health perception, physical health, physically-conditioned role function, physical pain, vitality, mental health, emotionally-related role function, social functionality. Different Likert-Scales are used. A physical sum scale and a psychological sum scale can be calculated. The polarity of four items must be reversed so that higher values in all items and total scales reflect a better state of health. Normative data are available. Values may range from 0-100, with a mean of 50 and a standard deviation of 10 in the general population. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Brief Symptom Inventory (BSI) | Within the first 7 days after admission
  Questionnaire on the burden of symptoms. The BSI is also called the Brief Symptom Check List (BSCL), it is a short form of the SCL-90 (Derogatis, 1993). The BSI consists of 53 items (physical as well as psychological symptoms), which are assessed subjectively on a Likert scale in relation to the last seven days from 0 = "not at all" to 5 = "very strong". The items result in nine scales: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.
Demographic data and chronic complaints and current illnesses | Within the first 7 days after admission
  Age, sex, height, weight, body mass index, and further demographic data. Chronic complaints and current illnesses.

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Clinic, Dept. of Physical Medicine & Rehabilitation, Linz, Austria

IPD SHARING:
Plan to Share IPD: No